CLINICAL TRIAL: NCT02614118
Title: Premedication Efficacy of Oral Ketorolac and Ketorolac/ Acetaminophen on Post Endodontic Treatment Pain
Brief Title: Premedication Efficacy of Oral Ketorolac and Ketorolac/ Acetaminophen on Post Treatment Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nahid Mohammadzadeh Akhlaghi, Associate Professor, Azad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AZadUMS-P/139/D
Record Dates: First submitted 2015-11-19; First posted 2015-11-25 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Irreversible Pulpitis
Keywords: Endodontic treatment; non steroid; pain; pre medication
MeSH Terms: conditions — Pain | interventions — Ketorolac Tromethamine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ketorolac tromethanine (Active Comparator): 10 mg oral Ketorolac tromethanine 45 minutes before root canal treatment
  Interventions: Drug: Ketorolac tromethamine
- Acetaminphen & Ketorolac tromethamine (Active Comparator): 1000 mg Acetaminophen and 10 mg Ketorolac tromethamine oral 45 minutes before root canal treatment
  Interventions: Drug: Ketorolac tromethamine; Drug: Acetaminophen
- Placebo (Placebo Comparator): placebo 45 minutes before root canal treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac tromethamine — 10 mg oral Ketorolac tromethamine 45 minutes before root canal treatment
  Other Names: Toradol
  Arms: Acetaminphen & Ketorolac tromethamine; Ketorolac tromethanine
Drug: Acetaminophen — 1000 mg oral Acetaminophen along with10 mg oral Ketorolac tromethamine 45 minutes before root canal treatment.
  Other Names: Tylenol
  Arms: Acetaminphen & Ketorolac tromethamine
Drug: Placebo — placebo 45 minutes before root canal treatment
  Other Names: disambiguation
  Arms: Placebo

SUMMARY:
The aim of this study is premedication efficacy of analgesics on post endodontic pain. Sixty-six healthy adult volunteers including criteria, are participating. The patients will be divided into 3 groups and will be randomly given one of pre medications including 1) 10 mg Ketorolac, 2) 10 mg Ketorolac plus 1000mg Acetaminophen, and 3)Placebo, 45 minutes before applying the injection. All patients will receive standard root canal treatment. Patients will record their post treatment pain using a Heft parker Visual Analog Scale(VAS). Success will be considered as no or mild pain (VAS≤54)with no need to take analgesic. Data will be analysed using Mann-U-Whitney and Kruskal-wallis tests.

DETAILED DESCRIPTION:
The aim of this study is premedication efficacy of analgesics on post endodontic pain. Sixty-six healthy adult volunteers with age ranged 18-65, non smoking or any medicine consumption, non pregnant or break feeding who haven't received any analgesic during 24 hours before the treatment, are participating. The patients will be divided into 3 groups and will be randomly given one of premedications including 1) 10 mg Ketorolac, 2) 10 mg Ketorolac plus 1000mg Acetaminophen, and 3)Placebo, 45 minutes before the treatment. All patients will receive a standard root canal treatment. Patients will record their post treatment pain using a Heft parker Visual Analog Scale(VAS). Success will be considered as no or mild pain (VAS≤54) with no need to take analgesic during 6, 12, 24 and 48 hours intervals following the treatment. Data will be analysed using Mann-U-Whitney and Kruskal-wallis tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ranged 18-65
* without systemic diseases
* without any medicine consumption
* non smoking
* non pregnant
* non breast feeding
* with asymptomatic irreversible pulpitis ( Visual Analog Scale ≤ 54) in one mandibular molar that needs root canal treatment
* without any medicine consumption or analgesic and sedation who understand and sign the VAS and consent forms.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pain rate change based on visual analog scale(VAS) form | 6,12,24,and 48 hour intervals
  Each patient receives a VAS form and record his/her pain rate on the VAS form whenever he/she feels any pain during each interval after the treatment. If the patient has to take any analgesic, she/he will record the pain rate on that interval and will not continue filling the forms out on the next intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Nahid Mohammadzadeh Akhlaghi, DDS,MDS, Principal Investigator — Associate Professor
Locations (1):
- Dental Branch, AZad UMS, Tehran, Tehran Province, Iran